CLINICAL TRIAL: NCT00869245
Title: Efficacy Evaluation of Observation Unit Cardiac Magnetic Resonance Imaging (MRI) in Patients With Intermediate Risk Acute Chest Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00008247; AHA Identification # 0980008N
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-04

CONDITIONS: Acute Coronary Syndrome; Chest Pain
Keywords: ACS; Acute Coronary Syndrome; Chest pain; Cardiac MRI; CMR; Risk Stratification; Emergency Department
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Emergencies

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Cardiac MRI Protocol. Patients will be transferred to the observation unit and undergo a stress cardiac MRI evaluation.
  Interventions: Other: OU - Cardiac MRI
- 2 (Experimental): Conventional care cardiac testing. Patients will be transferred to the observation unit and undergo cardiac testing as determined by their treating physician.
  Interventions: Other: OU - Conventional Care Testing

INTERVENTIONS:
Other: OU - Cardiac MRI — During ED evaluation, patients are randomized to cardiac MRI or conventional care testing.
  Arms: 1
Other: OU - Conventional Care Testing — Patients in the conventional testing arm will undergo testing as determined by their treating physician.
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the best way to evaluate patients with chest pain in the emergency department. It compares types of cardiac tests performed while receiving treatment in an observation unit. Patients will either undergo cardiac MRI testing or conventional care testing. Patients treated in the conventional care testing group will undergo the testing their doctor determines is best for them. All patients will undergo follow up to find out if they have had any heart related events.

DETAILED DESCRIPTION:
Despite spending $12 billion annually on the emergency evaluation of chest pain in the US, only 15% of admitted patients have a cardiac cause of their presenting symptoms. Observation units (OU) improve resource utilization, are endorsed by the ACC/AHA guidelines, but have seen limited implementation in non-low risk chest pain patients due to limitations of traditional cardiac testing. Cardiac magnetic resonance imaging (CMR) is sensitive and specific for ischemia, can simultaneously assess cardiac function and myocardial perfusion, and could revolutionize the diagnostic process for intermediate risk patients with chest pain. The superior accuracy of CMR could decrease testing resulting from false positive results. The high sensitivity for ongoing ischemia could allow imaging in parallel with cardiac markers.

Research hypotheses:

OU-CMR will have superior therapeutic efficacy to OU-conventional testing.

An OU-CMR strategy will have higher diagnostic thinking efficacy than OU-conventional testing.

Methods summary:

To address the question of feasibility of a CMR approach to managing patients at intermediate risk for ACS, we propose a randomized clinical trial of 120 patients at intermediate risk of ACS that present to the ED of Wake Forest University Baptist Medical Center (WFUBMC) for evaluation of chest pain. All patients will receive care in an OU, and will be randomized to CMR, or conventional testing. CMR participants will undergo cardiac markers and CMR testing; conventional testing participants will undergo serial cardiac markers followed by conventional cardiac testing. ACS (infarction, death, coronary revascularization, unstable angina) will be assessed by evaluation of hospital course and phone follow-up at 30 days. Cost of hospital care will be compared among groups.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Chest discomfort or other symptoms consistent with possible ACS
* TIMI risk score ≥ 1 or physician impression* of intermediate or high likelihood symptoms represent ACS
* Patient requires an inpatient or observation unit evaluation for their chest pain
* The treating physician feels the patient could be discharged home if cardiac disease was excluded
* ED attending feels patient is safe for observation unit care**

Exclusion Criteria:

* Initial troponin I > 1.0 ng/ml
* New ST-segment elevation (≥1mV) or depression (≥2 mV)
* Contra-indications to MRI (listed below)
* Unable to lie flat
* Hypotension (systolic < 90 mm Hg)
* Renal insufficiency (estimated GFR < 45 cc/min) or end stage renal disease
* Life expectancy less than 3 months
* Patient refusal of medical record review and follow-up at 30 days
* Pregnancy
* Liver, heart, or kidney transplant
* Chronic liver disease
* Unable to speak English or Spanish
* The ED attending feels that cardiac catheterization is indicated
* The ED care provider intends to order a CT coronary angiogram

(*)Physicians are encouraged to use the 2007 ACC/AHA guidelines for the management of patients with NSTE ACS as a framework for this assessment.(1)

(**)These patients should generally not be considered for observation unit care: PCI / CAGB in past 6 months, multiple stents, multiple prior MIs

Contraindications to MRI: (Pacemaker, defibrillator, cerebral aneurysm clips, metallic ocular foreign body, implanted devices, claustrophobia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Therapeutic efficacy: Length of stay | Duration of Initial Hospitalization

SECONDARY OUTCOMES:
Therapeutic efficacy: Correct cardiovascular admission decision | Duration of Initial Hospitalization
Therapeutic efficacy: Non-therapeutic cardiac catheterizations | 30 days
Diagnostic thinking efficacy: change in diagnostic certainty | 30 days
Cost of index hospitalization | Duration of Initial Hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Miller, M.D., Principal Investigator — WFUBMC
Locations (1):
- Wake Forest University Baptist Medical Center - Emergency Department, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr, Jacobs AK, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction); American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Academic Emergency Medicine. ACC/AHA 2007 guidelines for the management of patients with unstable angina/non ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction): developed in collaboration with the American College of Emergency Physicians, the Society for Cardiovascular Angiography and Interventions, and the Society of Thoracic Surgeons: endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic Emergency Medicine. Circulation. 2007 Aug 14;116(7):e148-304. doi: 10.1161/CIRCULATIONAHA.107.181940. Epub 2007 Aug 6. No abstract available. PMID 17679616
- [Background] Rosamond W, Flegal K, Friday G, Furie K, Go A, Greenlund K, Haase N, Ho M, Howard V, Kissela B, Kittner S, Lloyd-Jones D, McDermott M, Meigs J, Moy C, Nichol G, O'Donnell CJ, Roger V, Rumsfeld J, Sorlie P, Steinberger J, Thom T, Wasserthiel-Smoller S, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2007 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2007 Feb 6;115(5):e69-171. doi: 10.1161/CIRCULATIONAHA.106.179918. Epub 2006 Dec 28. No abstract available. PMID 17194875
- [Background] McCaig LF, Nawar EW. National Hospital Ambulatory Medical Care Survey: 2004 emergency department summary. Adv Data. 2006 Jun 23;(372):1-29. PMID 16841785
- [Background] Christenson J, Innes G, McKnight D, Thompson CR, Wong H, Yu E, Boychuk B, Grafstein E, Rosenberg F, Gin K, Anis A, Singer J. A clinical prediction rule for early discharge of patients with chest pain. Ann Emerg Med. 2006 Jan;47(1):1-10. doi: 10.1016/j.annemergmed.2005.08.007. Epub 2005 Oct 19. PMID 16387209
- [Background] Goldstein JA, Gallagher MJ, O'Neill WW, Ross MA, O'Neil BJ, Raff GL. A randomized controlled trial of multi-slice coronary computed tomography for evaluation of acute chest pain. J Am Coll Cardiol. 2007 Feb 27;49(8):863-71. doi: 10.1016/j.jacc.2006.08.064. Epub 2007 Feb 12. PMID 17320744
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Background] Heller GV, Stowers SA, Hendel RC, Herman SD, Daher E, Ahlberg AW, Baron JM, Mendes de Leon CF, Rizzo JA, Wackers FJ. Clinical value of acute rest technetium-99m tetrofosmin tomographic myocardial perfusion imaging in patients with acute chest pain and nondiagnostic electrocardiograms. J Am Coll Cardiol. 1998 Apr;31(5):1011-7. doi: 10.1016/s0735-1097(98)00057-6. PMID 9562001
- [Background] Sprivulis PC, Da Silva JA, Jacobs IG, Frazer AR, Jelinek GA. The association between hospital overcrowding and mortality among patients admitted via Western Australian emergency departments. Med J Aust. 2006 Mar 6;184(5):208-12. doi: 10.5694/j.1326-5377.2006.tb00416.x. PMID 16515429
- [Background] Miro O, Antonio MT, Jimenez S, De Dios A, Sanchez M, Borras A, Milla J. Decreased health care quality associated with emergency department overcrowding. Eur J Emerg Med. 1999 Jun;6(2):105-7. doi: 10.1097/00063110-199906000-00003. PMID 10461551
- [Background] Pope JH, Aufderheide TP, Ruthazer R, Woolard RH, Feldman JA, Beshansky JR, Griffith JL, Selker HP. Missed diagnoses of acute cardiac ischemia in the emergency department. N Engl J Med. 2000 Apr 20;342(16):1163-70. doi: 10.1056/NEJM200004203421603. PMID 10770981
- [Background] Braunwald E, Antman EM, Beasley JW, Califf RM, Cheitlin MD, Hochman JS, Jones RH, Kereiakes D, Kupersmith J, Levin TN, Pepine CJ, Schaeffer JW, Smith EE 3rd, Steward DE, Theroux P, Gibbons RJ, Alpert JS, Faxon DP, Fuster V, Gregoratos G, Hiratzka LF, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association. Committee on the Management of Patients With Unstable Angina. ACC/AHA 2002 guideline update for the management of patients with unstable angina and non-ST-segment elevation myocardial infarction--summary article: a report of the American College of Cardiology/American Heart Association task force on practice guidelines (Committee on the Management of Patients With Unstable Angina). J Am Coll Cardiol. 2002 Oct 2;40(7):1366-74. doi: 10.1016/s0735-1097(02)02336-7. No abstract available. PMID 12383588
- [Background] Hoffmann U, Nagurney JT, Moselewski F, Pena A, Ferencik M, Chae CU, Cury RC, Butler J, Abbara S, Brown DF, Manini A, Nichols JH, Achenbach S, Brady TJ. Coronary multidetector computed tomography in the assessment of patients with acute chest pain. Circulation. 2006 Nov 21;114(21):2251-60. doi: 10.1161/CIRCULATIONAHA.106.634808. Epub 2006 Oct 30. PMID 17075011
- [Background] Hollander JE, Litt HI, Chase M, Brown AM, Kim W, Baxt WG. Computed tomography coronary angiography for rapid disposition of low-risk emergency department patients with chest pain syndromes. Acad Emerg Med. 2007 Feb;14(2):112-6. doi: 10.1197/j.aem.2006.09.051. PMID 17267528
- [Background] Katz DA, Griffith JL, Beshansky JR, Selker HP. The use of empiric clinical data in the evaluation of practice guidelines for unstable angina. JAMA. 1996 Nov 20;276(19):1568-74. PMID 8918854
- [Background] Gomberg-Maitland M, Murphy SA, Moliterno DJ, Cannon CP. Are we appropriately triaging patients with unstable angina? Am Heart J. 2005 Apr;149(4):613-8. doi: 10.1016/j.ahj.2004.09.035. PMID 15990742
- [Background] Stowers SA, Eisenstein EL, Th Wackers FJ, Berman DS, Blackshear JL, Jones AD Jr, Szymanski TJ Jr, Lam LC, Simons TA, Natale D, Paige KA, Wagner GS. An economic analysis of an aggressive diagnostic strategy with single photon emission computed tomography myocardial perfusion imaging and early exercise stress testing in emergency department patients who present with chest pain but nondiagnostic electrocardiograms: results from a randomized trial. Ann Emerg Med. 2000 Jan;35(1):17-25. doi: 10.1016/S0196-0644(00)70100-4. PMID 10613936
- [Background] Tatum JL, Jesse RL, Kontos MC, Nicholson CS, Schmidt KL, Roberts CS, Ornato JP. Comprehensive strategy for the evaluation and triage of the chest pain patient. Ann Emerg Med. 1997 Jan;29(1):116-25. doi: 10.1016/s0196-0644(97)70317-2. PMID 8998090
- [Background] Bashore TM, Bates ER, Berger PB, Clark DA, Cusma JT, Dehmer GJ, Kern MJ, Laskey WK, O'Laughlin MP, Oesterle S, Popma JJ, O'Rourke RA, Abrams J, Bates ER, Brodie BR, Douglas PS, Gregoratos G, Hlatky MA, Hochman JS, Kaul S, Tracy CM, Waters DD, Winters WL Jr; American College of Cardiology. Task Force on Clinical Expert Consensus Documents. American College of Cardiology/Society for Cardiac Angiography and Interventions Clinical Expert Consensus Document on cardiac catheterization laboratory standards. A report of the American College of Cardiology Task Force on Clinical Expert Consensus Documents. J Am Coll Cardiol. 2001 Jun 15;37(8):2170-214. doi: 10.1016/s0735-1097(01)01346-8. No abstract available. PMID 11419904
- [Background] Desai AS, Solomon DH, Stone PH, Avorn J. Economic consequences of routine coronary angiography in low- and intermediate-risk patients with unstable angina pectoris. Am J Cardiol. 2003 Aug 15;92(4):363-7. doi: 10.1016/s0002-9149(03)00650-7. PMID 12914862
- [Background] Calvin JE, Klein LW, VandenBerg EJ, Meyer P, Parrillo JE. Validated risk stratification model accurately predicts low risk in patients with unstable angina. J Am Coll Cardiol. 2000 Nov 15;36(6):1803-8. doi: 10.1016/s0735-1097(00)00977-3. PMID 11092647
- [Background] Ramakrishna G, Milavetz JJ, Zinsmeister AR, Farkouh ME, Evans RW, Allison TG, Smars PA, Gibbons RJ. Effect of exercise treadmill testing and stress imaging on the triage of patients with chest pain: CHEER substudy. Mayo Clin Proc. 2005 Mar;80(3):322-9. doi: 10.4065/80.3.322. PMID 15757012
- [Background] Goodacre S, Cross E, Lewis C, Nicholl J, Capewell S; ESCAPE Research Team. Effectiveness and safety of chest pain assessment to prevent emergency admissions: ESCAPE cluster randomised trial. BMJ. 2007 Sep 29;335(7621):659. doi: 10.1136/bmj.39325.624109.AE. Epub 2007 Sep 18. PMID 17878265
- [Background] Kwong RY, Schussheim AE, Rekhraj S, Aletras AH, Geller N, Davis J, Christian TF, Balaban RS, Arai AE. Detecting acute coronary syndrome in the emergency department with cardiac magnetic resonance imaging. Circulation. 2003 Feb 4;107(4):531-7. doi: 10.1161/01.cir.0000047527.11221.29. PMID 12566362
- [Background] Abdel-Aty H, Zagrosek A, Schulz-Menger J, Taylor AJ, Messroghli D, Kumar A, Gross M, Dietz R, Friedrich MG. Delayed enhancement and T2-weighted cardiovascular magnetic resonance imaging differentiate acute from chronic myocardial infarction. Circulation. 2004 May 25;109(20):2411-6. doi: 10.1161/01.CIR.0000127428.10985.C6. Epub 2004 May 3. PMID 15123531
- [Background] Plein S, Greenwood JP, Ridgway JP, Cranny G, Ball SG, Sivananthan MU. Assessment of non-ST-segment elevation acute coronary syndromes with cardiac magnetic resonance imaging. J Am Coll Cardiol. 2004 Dec 7;44(11):2173-81. doi: 10.1016/j.jacc.2004.08.056. PMID 15582315
- [Background] Nagel E, Lehmkuhl HB, Bocksch W, Klein C, Vogel U, Frantz E, Ellmer A, Dreysse S, Fleck E. Noninvasive diagnosis of ischemia-induced wall motion abnormalities with the use of high-dose dobutamine stress MRI: comparison with dobutamine stress echocardiography. Circulation. 1999 Feb 16;99(6):763-70. doi: 10.1161/01.cir.99.6.763. PMID 9989961
- [Background] Fryback DG, Thornbury JR. The efficacy of diagnostic imaging. Med Decis Making. 1991 Apr-Jun;11(2):88-94. doi: 10.1177/0272989X9101100203. PMID 1907710
- [Background] Carlos R. Introduction to cost-effectiveness analysis in radiology: principles and practical application. Acad Radiol. 2004 Feb;11(2):141-8. doi: 10.1016/s1076-6332(03)00649-4. PMID 14974588
- [Background] Hollander JE, Blomkalns AL, Brogan GX, Diercks DB, Field JM, Garvey JL, Gibler WB, Henry TD, Hoekstra JW, Holroyd BR, Hong Y, Kirk JD, O'Neil BJ, Jackson RE; Multidisciplinary Standardized Reporting Criteria Task Force. Standardized reporting guidelines for studies evaluating risk stratification of ED patients with potential acute coronary syndromes. Acad Emerg Med. 2004 Dec;11(12):1331-40. doi: 10.1197/j.aem.2004.08.033. No abstract available. PMID 15576525
- [Background] Kline JA, Mitchell AM, Runyon MS, Jones AE, Webb WB. Electronic medical record review as a surrogate to telephone follow-up to establish outcome for diagnostic research studies in the emergency department. Acad Emerg Med. 2005 Nov;12(11):1127-33. doi: 10.1197/j.aem.2005.04.012. Epub 2005 Sep 15. PMID 16166598
- [Background] Tsushima Y, Aoki J, Endo K. Contribution of the diagnostic test to the physician's diagnostic thinking: new method to evaluate the effect. Acad Radiol. 2003 Jul;10(7):751-5. doi: 10.1016/s1076-6332(03)80120-4. PMID 12862284
- [Background] Puskas JD, Williams WH, Mahoney EM, Huber PR, Block PC, Duke PG, Staples JR, Glas KE, Marshall JJ, Leimbach ME, McCall SA, Petersen RJ, Bailey DE, Weintraub WS, Guyton RA. Off-pump vs conventional coronary artery bypass grafting: early and 1-year graft patency, cost, and quality-of-life outcomes: a randomized trial. JAMA. 2004 Apr 21;291(15):1841-9. doi: 10.1001/jama.291.15.1841. PMID 15100202
- [Background] Myocardial infarction redefined--a consensus document of The Joint European Society of Cardiology/American College of Cardiology Committee for the redefinition of myocardial infarction. Eur Heart J. 2000 Sep;21(18):1502-13. doi: 10.1053/euhj.2000.2305. PMID 10973764
- [Background] Miller CD, Fermann GJ, Lindsell CJ, Mahaffey KW, Peacock WF, Pollack CV, Hollander JE, Diercks DB, Gibler WB, Hoekstra JW; EMCREG-International itrACS Investigators. Initial risk stratification and presenting characteristics of patients with evolving myocardial infarctions. Emerg Med J. 2008 Aug;25(8):492-7. doi: 10.1136/emj.2007.052183. PMID 18660397
- [Background] Cury RC, Shash K, Nagurney JT, Rosito G, Shapiro MD, Nomura CH, Abbara S, Bamberg F, Ferencik M, Schmidt EJ, Brown DF, Hoffmann U, Brady TJ. Cardiac magnetic resonance with T2-weighted imaging improves detection of patients with acute coronary syndrome in the emergency department. Circulation. 2008 Aug 19;118(8):837-44. doi: 10.1161/CIRCULATIONAHA.107.740597. Epub 2008 Aug 4. PMID 18678772
- [Background] Mahaffey KW, Puma JA, Barbagelata NA, DiCarli MF, Leesar MA, Browne KF, Eisenberg PR, Bolli R, Casas AC, Molina-Viamonte V, Orlandi C, Blevins R, Gibbons RJ, Califf RM, Granger CB. Adenosine as an adjunct to thrombolytic therapy for acute myocardial infarction: results of a multicenter, randomized, placebo-controlled trial: the Acute Myocardial Infarction STudy of ADenosine (AMISTAD) trial. J Am Coll Cardiol. 1999 Nov 15;34(6):1711-20. doi: 10.1016/s0735-1097(99)00418-0. PMID 10577561
- [Background] Ross AM, Gibbons RJ, Stone GW, Kloner RA, Alexander RW; AMISTAD-II Investigators. A randomized, double-blinded, placebo-controlled multicenter trial of adenosine as an adjunct to reperfusion in the treatment of acute myocardial infarction (AMISTAD-II). J Am Coll Cardiol. 2005 Jun 7;45(11):1775-80. doi: 10.1016/j.jacc.2005.02.061. PMID 15936605
- [Background] Karha J, Gibson CM, Murphy SA, Dibattiste PM, Cannon CP; TIMI Study Group. Safety of stress testing during the evolution of unstable angina pectoris or non-ST-elevation myocardial infarction. Am J Cardiol. 2004 Dec 15;94(12):1537-9. doi: 10.1016/j.amjcard.2004.08.033. PMID 15589011
- [Background] Geleijnse ML, Elhendy A, Kasprzak JD, Rambaldi R, van Domburg RT, Cornel JH, Klootwijk AP, Fioretti PM, Roelandt JR, Simoons ML. Safety and prognostic value of early dobutamine-atropine stress echocardiography in patients with spontaneous chest pain and a non-diagnostic electrocardiogram. Eur Heart J. 2000 Mar;21(5):397-406. doi: 10.1053/euhj.1999.1860. PMID 10666354
- [Derived] Miller CD, Hoekstra JW, Lefebvre C, Blumstein H, Hamilton CA, Harper EN, Mahler S, Diercks DB, Neiberg R, Hundley WG. Provider-directed imaging stress testing reduces health care expenditures in lower-risk chest pain patients presenting to the emergency department. Circ Cardiovasc Imaging. 2012 Jan;5(1):111-8. doi: 10.1161/CIRCIMAGING.111.965293. Epub 2011 Nov 29. PMID 22128195